CLINICAL TRIAL: NCT01778777
Title: Safety, Function and Quality of Life in Patient With Rotator Cuff Tear Arthropathy Treated With the Univers® Revers Shoulder Prosthesis
Brief Title: Safety Study of Univers® Revers Shoulder Prosthesis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Schulthess Klinik (Other)
Collaborators: Arthrex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UniversRevers
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2023-04-18 (Actual); Status verified 2022-05

CONDITIONS: Rotator Cuff Tear Arthropathy
Keywords: rotator cuff tear arthropathy; inverse prosthesis; safety; universe reverse
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- UniverseReverse (Experimental): Cohort get an universe reverse prosthesis
  Interventions: Device: Universe Reverse Prosthesis

INTERVENTIONS:
Device: Universe Reverse Prosthesis — Implantation of an universe reverse prosthesis

SUMMARY:
The primary safety objective is to demonstrate that severe device-related complication (Serious Adverse Device Effect = SADE) occur within 2 years after prosthesis implantation at a rate of less than 2%. Such adverse events include (but are not limited to) revisions due to dislocation or glenoid loosening, septic arthritis and scapular fractures requiring surgical repair.

DETAILED DESCRIPTION:
Reverse shoulder arthroplasty and its principles are still recognized today as the gold standard for treatment of degenerative arthropathy of the shoulder associated with an irreparable tear of the rotator cuff. The new Arthrex Univers® Revers Shoulder Prosthesis shows a large and narrow range of components, whether it is a stem, cup, spacer, inlay or glenosphere. Adjustment can be done in very small steps to match anatomic and biomechanic needs. The Arthrex Univers Revers Shoulder Prosthesis is the only device up to date that can be configured in two different inclination angles without any limitation in component use.

This multicentre case-series has the goal to evaluate whether patients with rotator cuff tear arthropathy benefit from the Univers® Revers shoulder prosthesis in terms of low complication risk, as well as high function and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged 18 years and over
* Patient with primary omarthrosis or secondary osteoarthritis associated with insufficiency in the centering function of the rotator cuff

and

• Willing and able to give written informed consent to participate in the study including all follow-up examinations

Exclusion Criteria:

* Previous ipsilateral shoulder arthroplasty
* Acute shoulder trauma
* Post-traumatic secondary osteoarthritis
* Rheumatoid arthritis
* General medical contraindication to surgery
* Known hypersensitivity to the materials used
* Tumour / malignoma
* Any disease process that would preclude accurate evaluation (e.g. neuromuscular, psychiatric or metabolic disorder)
* Bacterial infection at the time point of operation
* Recent history of substance abuse
* Legal incompetence
* Pregnancy or
* Participation in any other medical device or medicinal product study within the previous months that could influence the results of the present study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2013-09-01 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2023-04-15 (Actual)

PRIMARY OUTCOMES:
SADE within 2 years po | 2 years po
  The primary safety objective is to demonstrate that severe device-related complication (Serious Adverse Device Effect = SADE) occur within 2 years after prosthesis implantation at a rate of less than 2%.

SECONDARY OUTCOMES:
Risk of adverse events intra-operatively, and post-operatively up to 2 years follow-up | 2 years
  As typically one single surgery should be sufficient to treat the patient, all secondary surgical interventions should be revisions due to a complication.
  The occurrence and time of revision surgery (implant survival) will be described by Kaplan-Meier curve.
Prosthesis survival at 2, 5 and 10 years | 2, 5 and 10 years
  All Patients with a prosthesis revision will be documented along with the date of revision. At each follow up time point the proportion of patients with prosthesis revision will be estimated. Time to prosthesis revision will be examined by survival methods to account for censored data.
Constant (Murley) score (CS) | 6mo, 1, 2, 5 and 10 years
  The Constant (Murley) score is possibly the most commonly used tool for assessment of shoulder function. The physician asks and documents answers to QOL questions (pain and ADL, ability to work, sleep, sports and leisure) and certain clinical parameters (active ROM, abduction strength). The different scales will be summed and normalized to O=worst to 100= best. A German version is available for clinical use. Investigators are obliged to use a spring balance for the force measurements. Only one measurement per patient per assessment will be done.
The Shoulder Pain and Disability Index (SPADI) | 6mo, 1, 2, 5 and 10 years
  The Shoulder Pain and Disability Index (SPADI) is a short, self-administered questionnaire that provides an item scoring by a visual analogue scale (VAS) from 0 (no pain/no difficulty, i.e. best) to 11 (worst pain imaginable/so difficult required help, i.e. worst). Five items assess pain and 8 items disability of the arm (function). The unweighted means of the 5 pain and the 8 function items will be transformed into the scale from 0 (=worst) to 100 (=best) for both scales and are used to determine pain and function scores. The average of these two scores then gives the total SPADI score. A validated German version is available.
Short version of the Disability of the Arm, Shoulder and Hand questionnaire (QuickDASH) | 6mo, 1, 2, 5 and 10 years
  The Disability of the Arm, Shoulder and Hand questionnaire (DASH) is a comprehensive self-administered questionnaire about symptoms and functioning of the entire upper extremity. The DASH enquires about the ability to perform simple and complex activities of daily living (ADL) that are commonly performed with either one or both arms. The total score is derived from the unweighted mean of 30 items, of which at least 27 have to be answered. The QuickDASH is a more efficient version of the DASH outcome measure that appears to retain its measurement properties. It contains eleven items and is similar with regard to scores and properties to the full DASH. A validated full-length German version is available that can be used in the shortened version.
EuroQoL EQ-5D-5L | 6wk, 6mo, 1, 2, 5 and 10 years
  The EQ-5D is a widely used instrument to measure and value generic health (status). It is based on a descriptive system that defines health in terms of 5 dimensions: Mobility, Self-Care, Usual Activities, Pain/Discomfort, and Anxiety/Depression. The instrument is designed for self-completion, and patients also rate their overall health on the day of the interview on a 0-100 visual analogue scale (EQ-VAS).
Patient satisfaction | 6wk, 6mo, 1, 2, 5 and 10 years
  In order to obtain an overall assessment of the arthroplasty result, patients will be asked to assess their current state of health in general related to the operated shoulder joint at the follow-up compared to the state before the arthroplasty. This so-called 'transition' question has the possible answers 'much worse', 'slightly worse', 'equal', 'slightly better', and 'much better'. Patients also rate their level of satisfaction, with the help of a numeric rating scale (NRS: 0-10), in terms of how the outcome met up to their preoperative expectations of the arthroplasty. Finally, they will be asked whether - with their current knowledge of the outcome - they would again choose the operation if they found themselves in similar circumstances to those which prevailed preoperatively.
Radiographic Parameters | 6mo, 1, 2, 5 and 10 years
  Three radiographs should be taken at each study visit: AP view in internal and external rotation and axial view. The images will be collected digitally and centralized for latter evaluation by an independent reviewer based on the radiographic assessment CRF developed by the Schulthess clinic, including the following parameters:
  * Scapular notching
  * Signs of osteolysis at the glenoid and at the stem
  * Status of tuberculum majus and minus
  * Glenoid migration
  * Glenoid component seating
  * Stem position
  * Change of relative position of components
  * Ectopic bone formation
  * Cortical bone resorption
  * Prosthesis breakage
  * Rotation failure
  * Luxation of the prosthesis
  * PE Wear of the metaglene
  * PE Dissociation
Patient active and passive range of motion (ROM) and shoulder strength | 6mo, 1, 2, 5 and 10 years
  The following active and passive range of motion parameters will be documented:
  * Abduction
  * Elevation
  * External rotation by 0°
  * External-internal rotation by 90°

CONTACTS AND LOCATIONS:
Overall Officials: Hans-Kaspar Schwyzer, Dr., Principal Investigator — Schulthess Klinik
Locations (1):
- Schulthess Klinik, Zurich, Canton of Zurich, Switzerland